CLINICAL TRIAL: NCT06888349
Title: The Effect of Combined IPACK(Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee) Block with Adductor Canal Block Versus Adductor Canal Block Alone on Pain Management and Early Mobility After Total Knee Arthroplasty
Brief Title: The Effect of Combined IPACK Block with ACB Versus ACB Alone on Pain Management and Early Mobility After Total Knee Arthroplasty
Acronym: IPACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esraa Alaa El Deen Mahmoud Abass, Esraa Alaa(Assistant lecturer at anesthesia,ICU and pain department of faculty of medicine/ Ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MD 19/2023
Record Dates: First submitted 2025-02-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain; Motor Activity
Keywords: Postoperative pain; Early rehabilitation
MeSH Terms: conditions — Pain, Postoperative; Motor Activity | interventions — Anesthesia, Spinal; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Masking Description: Arm1: received ultrasound guided adductor canal block (ACB) alone . Arm2:received ultrasound guided adductor canal block (ACB) as group A, in addition to ultrasound guided infiltration of the interspace between popliteal artery and the capsule of posterior knee (IPACK) block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- adductor canal block (ACB) alone (Active Comparator): received ultrasound guided adductor canal block (ACB) alone using 22 Gag spinal needle with injection of 15ml 0.25% bupivacaine with addition of 2mg dexamethasone and 2.5mcg /ml epinephrine as an adjuvant to prolong its action.
  Interventions: Procedure: spinal anesthesia; Procedure: Adductor Canal Block
- adductor canal block (ACB)in addition to (IPACK) block (Active Comparator): received ultrasound guided adductor canal block (ACB) as group A, in addition to ultrasound guided infiltration of the interspace between popliteal artery and the capsule of posterior knee (IPACK) block with either of the two previously mentioned approaches, using 22Gag spinal needle injecting 20ml 0.25%bupivacaine with addition of 2mg dexamethasone and 2.5mcg /ml epinephrine as an adjuvant to prolong its action.
  Interventions: Procedure: spinal anesthesia; Procedure: Adductor Canal Block; Procedure: interspace between Popliteal artery and capsule of knee (IPACK) block

INTERVENTIONS:
Procedure: spinal anesthesia — spinal anesthesia using 15 mg 0.5% hyperbaric bupivacaine in the sitting position at L3-4 or L4-5 intervertebral space.
Procedure: Adductor Canal Block — local anesthetic spread around the saphenous nerve in the adductor canal ultrasound guided using 22 Gag spinal needle with injection of 15ml 0.25% bupivacaine with addition of 2mg dexamethasone and 2.5mcg /ml epinephrine as an adjuvant to prolong its action.
Procedure: interspace between Popliteal artery and capsule of knee (IPACK) block — ultrasound guided Local anesthetic infiltration over the posterior aspect of the femur underneath the popliteal artery targeting the genicular nerves which are the articular branches of tibial and common peroneal nerves, posterior branches of the obturator nerve, and medial genicular nerve using 22Gag spinal needle injecting 20ml 0.25%bupivacaine with addition of 2mg dexamethasone and 2.5mcg /ml epinephrine as an adjuvant to prolong its action.
  Arms: adductor canal block (ACB)in addition to (IPACK) block

SUMMARY:
This trial was established to assess efficiency of IPACK block in combination with ACB in relieving postoperative pain , particularly posterior knee pain and providing early rehabilitation after TKA in comparison with ACB alone .

DETAILED DESCRIPTION:
This trial was established to assess efficiency of IPACK block in combination with ACB in relieving postoperative pain , particularly posterior knee pain and providing early rehabilitation after TKA in comparison with ACB alone .All patients were subjected to full history taking including current medications and thorough physical examination.

Age, sex, BMI and ASA physical status were recorded and Preoperative investigations were done to all patients including laboratory investigations as (complete blood picture, bleeding time, prothrombin time and activated partial thromboplastin time) and other investigations according to the patient's medical condition. The patients were fasting for 2 to 8 hours preoperatively. All patients were consented with a written consent for the spinal anesthesia and either of the peripheral regional blocks that were held after explaining the procedure. Intraoperatively, All patients were monitored by pulse oximeter, non-invasive blood pressure cuff and electrocardiogram for heart rate and rhythm. IV Access was applied. All patients received 0.03 mg/kg midazolam iv, granisetron 1mg iv and dexamethasone 10 mg iv as a prophylaxis against nausea and vomiting.Sign IN and Time OUT checklist were revised before starting the anesthetic procedure and the surgical procedure, respectively.All patients received spinal anesthesia using 15 mg 0.5% hyperbaric bupivacaine in the sitting position at L3-4 or L4-5 intervertebral space.All patients received Intraoperative fluids and sedation with intravenous dexmedetomidine if needed.Checking on the availability of intralipid (lipid emulsion 20%) nearby and preparation of the ultrasound device (investigators used in the recent study the Sonosite M-Turbo C Portable Ultrasound). After patients' stabilization, Patients were divided into 2 group.

Group A: received ultrasound guided adductor canal block (ACB) alone using 22 Gag spinal needle with injection of 15ml 0.25% bupivacaine with addition of 2mg dexamethasone and 2.5mcg /ml epinephrine as an adjuvant to prolong its action.

Group B: received ultrasound guided adductor canal block (ACB) as group A, in addition to ultrasound guided infiltration of the interspace between popliteal artery and the capsule of posterior knee (IPACK) block with either of the two previously mentioned approaches, using 22Gag spinal needle injecting 20ml 0.25%bupivacaine with addition of 2mg dexamethasone and 2.5mcg /ml epinephrine as an adjuvant to prolong its action. Postoperatively,All patients were transferred to the post anesthesia care unit (PACU).

All patients were monitored at (PACU) for oxygen saturation, heart rate and blood pressure for 2hours observational period.The two groups of patients were evaluated and compared as regard:

Degree of postoperative pain using Numerical Rating Scale (NRS) at the first 48 hrs. The first need for analgesic rescue (NRS score ≥ 4 [0: no pain 10: very severe pain]) at 2, 4, 6, 8, 12, 24, and 48 hr. and the total amount of analgesic rescues was determined. Analgesic rescue was provided using 1 gram paracetamol IV and 30mg ketorolac IV, while in a few cases titration of pethidine was used after failure of the determined analgesic rescue with paracetamol and ketorolac to provide pain relief.

The recovery of spinal motor blockade and early motor ability using Bromage score and the incidence of peroneal motor weakness (dorsiflexion of the ankle and toes).

Length of hospital stays (defined as the days from the end of surgery until discharge).

The first mobilization time recorded in hours. The Timed Up and Go (TUG)test (measured in seconds).This test was performed on the 1st and 2nd postoperative days.Postoperative 1st and 2nd-day Rang of Movement (ROM) measurements.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Patients of either sex
* Age: between 45 and 75 years.
* Physical status: ASA I- III.
* Weight: BMI between 28-40 kg/m2.
* Lesion: any patient with knee pathology requiring total knee arthroplasty (TKA)

Exclusion Criteria:

* o Body mass index >40 kg/m2.

  * ASA>III.
  * Patient's refusal.
  * Revision knee arthroplasty
  * Bilateral knee arthroplasty.
  * Lack of mental ability to provide informed consent.
  * Neuropathic pain or sensory disorders of the surgical limb.
  * Contraindication to regional anesthesia (intolerance to the study drugs, bleeding diathesis, coagulopathy, malignancy or infection at the site of block).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
postoperative pain degree | 48hours
  two groups of patients were evaluated and compared as regard the Degree of postoperative pain using Numerical Rating Scale (NRS) which consist of a series of numbers rating pain intensity, typically from 0 to 10 with 0 being "no pain" and 10 being "the worst pain imaginable.", So that the higher the number the worse is the pain . The numerical rating scale is recorded each 4hours at the first 48 hours.
The first time to need analgesic rescue . | 2days
  The first time to need analgesic rescue when (Numerical rating scale score
  ≥ 4 which means moderate to severe pain ) is recorded in hours (the Numerical rating scale consist of a series of numbers rating pain intensity, typically from 0 to 10 with 0 being "no pain" 1to3 being "mild pain,4to6 being "moderate pain "and 7to10 being "sever pain" . So that the higher the number the worse is the pain.
the total amount of analgesic rescues needed measured in numbers | 2days
  Number of analgesic rescues needed when patient's pain is moderate to sever

SECONDARY OUTCOMES:
Sex influence on degree of pain | At the time of patients' enrollment in the study.
  Two groups were compared as regard number of males and females in each group
Age | At the time of patients' enrollment in the study.
  The ages of patients in each group were recoded and compared .
BMI(kg/m2) | At the time of patients'enrollment in the study.
  BMI of each patient was recorded and the two groups were compared .
Motor recovery | 2days
  Motor recovery after spinal anesthesia blockade Determined by Bromage score done using clinical assessment of motor ability . Bromage a score is score of four levels where score 1 = free movement of legs and feet; score 2 = just able to flex knees with free movement of feet; score 3 = unable to flex knees, but with free movement of feet; and score 4 = unable to move legs or feet.so that score 4 means no motor recovery with complete motor blockade and a(the minimum value) and score 1 means complete motor recovery with no blockade (the maximum value)
Mobility recovery | 2days
  Timed up and go test is done for each patient assessing the ability and the time it takes the patient to move up from a chair and wake for three meters then get back to the chair and is recorded in seconds .
Degree of motor recovery | 2days
  Range of motion test is done for each patient assessing the extension and flexion ability of the knee with measuring and recording the degree of angle in between .
Fast recovery and early hospital discharge | 48hours
  Duration of hospital stay is recorded in hours for each patient , so that the patient with hospital stay duration beyond 48hours is considered of delayed rehabilitation and prolonged hospital stay .

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No